CLINICAL TRIAL: NCT01602497
Title: A Sham-controlled Trial of Effect of High-frequency Transcranial Magnetic Stimulation in the Management of Borderline Personality Disorder Patients
Brief Title: Trial of Effect of High-frequency Transcranial Magnetic Stimulation in the Management of Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 90-01-30-13200
Record Dates: First submitted 2012-05-16; First posted 2012-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline personality disorder; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS intervention group (Active Comparator): The rTMS intervention group undergo ten session of real TMS therapy.
  Interventions: Device: rTMS
- Sham group (Placebo Comparator): Patients will undergo ten session of sham rTMS.
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: rTMS — Patients undergone 10 session of high-frequency rTMS therapy over their left DLPFC
  Other Names: repetitive transcranial magnetic stimulation
  Arms: rTMS intervention group
Device: sham rTMS — Patients will undergo ten session of sham rTMS.
  Other Names: sham repetitive transcranial magnetic stimulation
  Arms: Sham group

SUMMARY:
This study is going to evaluate the effects of repetitive transcranial magnetic stimulation (rTMS) on Borderline Personality Disorder patients symptoms.

DETAILED DESCRIPTION:
There is a great body of literature about the positive effects of rTMS therapy on various psychiatric disorders. In this study we are going to evaluate the effects of high-frequency rTMS over the left dorsolateral prefrontal cortex (DLPFC)region in borderline personality disorder (BPD) patients. patients will be assessed by subjective measures for BPD.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed borderline personality disorder according to DSM IV.

Exclusion Criteria:

* Epilepsy
* Any metal device
* Psychotic disorders
* Bipolar mood disorder type 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Patients' reports | Change from baseline to two weeks
  changes in subjective measures from baseline to tenth day of treatment

SECONDARY OUTCOMES:
patient's report | Change from baseline to 1 month
  change in subjective measures from baseline to 1 month after treatment
Patient's report | Change from baseline to 3 month
  change in subjective measures form baseline to 3 month after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Arbabi, M.D., Study Director — Tehran University of Medical Sciences